CLINICAL TRIAL: NCT06507839
Title: A First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study To Assess the Safety, Tolerability, Pharmacokinetics, and Food Effect of Thrv-1268 in Healthy Adult Subjects
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetic of Thrv-1268
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thryv Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0269
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
Keywords: THRV-1268; Atrial Fibrillation; Serum glucocorticoid regulated kinase-1; SGK-1 inhibitor
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Single Ascending Dose (SAD) THRV-1268 (Experimental): 5 dosing cohorts will receive a single oral dose of THRV-1268. The highest dose of THRV-1268 to be administered is 500 mg.
  Interventions: Drug: THRV-1268
- Food Effect THRV-1268 (Experimental): food effect will be integrated into one of the SAD cohorts as a single dose, two-period with at least a 7-day washout, crossover cohort.
  Interventions: Drug: THRV-1268
- Multiple Ascending Dose (MAD) THRV-1268 (Experimental): 3 dosing cohorts will receive THRV-1268 in the morning on Day 1 to Day 7.
  Interventions: Drug: THRV-1268
- Single Ascending Dose (SAD) Placebo (Placebo Comparator): 5 dosing cohorts will receive a single oral dose of placebo.
  Interventions: Other: Placebo
- Food Effect Placebo (Placebo Comparator): Food effect will be integrated into one of the SAD cohorts as a single dose, two-period with at least a 7-day washout, crossover cohort.
  Interventions: Other: Placebo
- Multiple Ascending Dose (MAD) Placebo (Placebo Comparator): 3 dosing cohorts will receive placebo in the morning from Day 1 to Day 7.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: THRV-1268 — THRV-1268 a serum glucocorticoid regulated kinase 1 (SGK-1) inhibitor
  Arms: Food Effect THRV-1268; Multiple Ascending Dose (MAD) THRV-1268; Single Ascending Dose (SAD) THRV-1268
Other: Placebo — Matching placebo
  Arms: Food Effect Placebo; Multiple Ascending Dose (MAD) Placebo; Single Ascending Dose (SAD) Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled study to be conducted in 2 parts: single ascending dose (SAD) incorporating a food effect arm and multiple ascending dose (MAD). Potential participants for each part will undergo screening procedures within 28 days of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1.Provision of signed and dated Informed Consent Form (ICF). 2.Stated willingness to comply with all study procedures and availability for the duration of the study.

3.Healthy adult male or female subjects. 4.If female, meets one of the following criteria:

* Women of childbearing potential who agrees to use any of the acceptable contraceptive methods:

  1. Abstinence from heterosexual intercourse from Screening through at least 30 days from last study dose.
  2. One of the following highly-effective contraception methods:

     1. systemic contraceptives (combined birth control pills, injectable/implant/ insertable hormonal birth control products, or transdermal patch) used from at least 28 days prior to Screening through to at least 30 days from last study dose
     2. intrauterine device (with or without hormones) used from at least 28 days prior to Screening through to at least 30 days from last study dose
     3. male partner vasectomized at least 6 months prior to Screening visit
  3. One of the following double-barrier contraception methods used from Screening through at least 30 days from last study dose

     1. Male condom used simultaneously with diaphragm plus spermicide
     2. Male condom used simultaneously with cervical cap plus spermicide Or
* Physiological postmenopausal status, defined as the absence of menses for at least 12 months following cessation of all exogenous hormonal treatments (without an alternative medical condition) at Screening and prior to the first study drug administration and have follicle stimulating hormone (FSH) levels ≥ 40 mIU/mL at Screening (If subject is postmenopausal and has an FSH of < 40 mIU/mL, but meets all other criteria in (1) or (2) above as well as all the other inclusion criteria, screening estradiol serum level must be equal to or below 150 pmol/L. In the case of hysterectomy, if FSH and estradiol do not meet the criteria, eligibility for study participation will be based on medical judgment.).

Or

* Surgically sterile, defined as those who have had hysterectomy, bilateral oophorectomy and/or bilateral salpingectomy, or bilateral tubal ligation.

  5.Men who are biologically capable of fathering children must agree and commit to use an adequate form of contraception (see female criteria 3) for the duration of the treatment period and for no less than 90 days after the last study dose. A male subject is considered capable of fathering children even if his sexual partner is sterile or using contraceptives.

  6.Men who are biologically capable of fathering children must also agree to refrain from sperm donation for the duration of the treatment period and for at least 90 days after the last study dose.

  7.Aged at least 18 years but not older than 60 years (inclusive). 8.Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively. 9.Non- or ex-smoker (An ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration).

  10.Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings in the physical examination (including vital signs) and/or ECG, as determined by an Investigator.

Exclusion Criteria:

1. Clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition, which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Clinically significant abnormal findings on the physical examination or medical history during Screening as deemed by the Investigator.
3. Female who is lactating.
4. Female who is pregnant according to the pregnancy test at Screening or prior to the first study drug administration.
5. Male subjects with a history of oligospermia or azoospermia or any other disorder of the reproductive system.
6. Male subjects who are undergoing treatment or evaluation for infertility.
7. The average of 3 measurements performed approximately 5 min apart: Screening or baseline (Day -1) diastolic BP <50 mmHg or >95; systolic BP <100 mmHg or >145 mmHg; or HR ≤ 50 beats per minute (bpm) using a validated digital BP device. These can be repeated in triplicate once after an additional quiet resting period.
8. Orthostatic BP performed after sitting quietly for at least 4 minutes and then standing for 2 minutes with a duplicate set performed after at least 3 minutes of sitting, with a reduction in systolic BP >20 mmHg, a reduction in diastolic BP >10 mmHg, or an increase in HR >20 bpm using a validated digital BP device.
9. Estimated creatinine clearance < 80 mL/min at Screening.
10. History of significant hypersensitivity to THRV-1268, kinase inhibitors or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
11. Screening 12-lead ECG demonstrating at least one of the following: PR >220 ms; QRS >110 ms, or QTcF >440 ms; atrioventricular block; branch bundle block, significant ST-T wave abnormalities or flat T waves that could interfere with QT analysis. Heart rate ≤50 bpm or >100 bpm.
12. History or evidence of any of the following: myocardial infarction; cardiac valvulopathy; cardiac surgery revascularization (coronary artery bypass grafting or percutaneous, transluminal coronary angioplasty); unstable angina; cerebrovascular accident, stroke, or transient ischemic attack; pacemaker; AF, flutter, or nonsustained or sustained ventricular tachycardia; orthostatic hypotension or orthostatic dizziness or lightheadedness, pulmonary arterial hypertension; sick sinus syndrome, second- or third-degree atrioventricular block; uncontrolled hypertension; congestive heart failure; personal or family history of sudden death or long QT syndrome; unexplained syncope or syncope within the last 3 years regardless of etiology.
13. Immunization with a Coronavirus Disease (COVID-19) vaccine in the 14 days prior to the first study drug administration.
14. Scheduled immunization with a COVID-19 vaccine during the study that, in the opinion of an Investigator, could potentially interfere with subject participation, subject safety, study results, or any other reason.
15. Use of immunosuppressant in the 28 days or 5 half-lives (whichever is longer) prior to the first study drug administration.
16. Major surgery with prolonged immobilization in the 28 days prior to the first study drug administration.
17. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic).
18. Any clinically significant illness in the 28 days prior to the first study drug administration.
19. Use of any over-the-counter or nutritional supplements in the last 7 days prior to the first study drug administration and during the study, that in the opinion of an Investigator would put into question the status of the subject as healthy.
20. Use of any prescription drugs (except for hormonal contraceptives or hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of an Investigator would put into question the status of the subject as healthy.
21. Use of St. John's wort in the 28 days prior to the first study drug administration.
22. Any history of tuberculosis.
23. Hemoglobin value below the lower limit of the reference laboratory at Screening, unless deemed non-significant by the Investigator.
24. Abnormal screening values in potassium, magnesium, alanine transaminase (ALT), aspartate aminotransferase, gamma-glutamyl transferase, alkaline phosphatase, total bilirubin, and direct bilirubin values, unless deemed non-significant by the Investigator.
25. Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first drug administration.
26. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus antibody tests.
27. Any other clinically significant abnormalities in laboratory test results at Screening that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
28. History of prior administration of THRV-1268 or inclusion in a previous cohort for this clinical study.
29. Intake of an IP or participation in a clinical trial in the 28 days or 5 half-lives (whichever is longer) prior to the first study drug administration.
30. Unable or unwilling to adhere to the lifestyle and dietary requirements described in Section 4.4.
31. Special diet or substantial changes in eating habits in the last 1 month before Screening.
32. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration.
33. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Number of Participants with Adverse Events | SAD: Day 7; Food Effect: Day 15; MAD: Day 16
  Number of Participants with Adverse Events

SECONDARY OUTCOMES:
Pharmacokinetic LQT-1268 AUC0-t | SAD: Day 1; Food Effect: Serially on Day 1 and Day 8; MAD: Serially on Day 1 and 7
  Area under the concentration-time curve (AUC) from time 0 to the time of the last
Pharmacokinetic LQT-1268 Cmax | SAD: Day 1; Food Effect: Serially on Day 1 and Day 8; MAD: Serially on Day 1 and 7
  Maximum observed plasma drug concentration
Pharmacokinetic LQT-1268 Tmax | SAD: Day 1; Food Effect: Serially on Day 1 and Day 8; MAD: Serially on Day 1 and 7
  Time to maximum observed plasma drug concentration
Pharmacokinetic LQT-1268 t1/2 | SAD: Day 1; Food Effect: Serially on Day 1 and Day 8; MAD: Serially on Day 1 and 7
  Time to maximum observed plasma drug concentration
Urine Pharmacokinetics of LQT-1268: Ae | SAD: Day 1; MAD: Serially on Day 1 and 7
  Amount of the administered dose recovered over the entire 24-hour interval
Urine Pharmacokinetics of LQT-1268: Fe | SAD: Day 1; MAD: Serially on Day 1 and 7
  Percentage of the administered dose recovered over the entire 24-hour interval
Urine Pharmacokinetics of LQT-1268: Ae0-t | SAD: Day 1; MAD: Serially on Day 1 and 7
  Amount excreted unchanged in urine over a given time interval
Plasma Pharmacokinetics of LQT-1268: Ctrough | MAD: Days 3-6
  Concentration of drug in the blood immediately before the next dose is administered
Plasma Pharmacokinetics of LQT-1268: Rac(AUC) | MAD: Day 7
  Drug accumulation ratio
Plasma Pharmacokinetics of LQT-1268: Rac(Cmax) | MAD: Day 7
  Drug accumulation ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences, Montreal, Quebec, Canada